CLINICAL TRIAL: NCT01792297
Title: The Effect of Bovine Colostrum Supplementation in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Principal Investigator, Phil Chilibeck, Ph.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12-255
Record Dates: First submitted 2013-02-04; First posted 2013-02-15 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Sarcopenia; Osteoporosis
Keywords: Sarcopenia; Osteoporosis; Cognition; Inflammation
MeSH Terms: conditions — Sarcopenia; Osteoporosis; Inflammation | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bovine Colostrum (Experimental): 60 g/d bovine colostrum in powder form to be mixed with drinks. The dose will be spread out 3 times per day (20 g per dose)
  Interventions: Dietary Supplement: Bovine colostrum
- Whey protein (Active Comparator): 60 g/d whey protein powder mixed into drinks. It is to be divided into 3 daily doses (20 g per dose)
  Interventions: Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Bovine colostrum
  Arms: Bovine Colostrum
Dietary Supplement: Whey protein
  Arms: Whey protein

SUMMARY:
Bovine colostrum is the initial milk secreted by cows during the first day after calving. Colostrum is high in protein and contains a number of substances that have potential to be beneficial for the immune system. Preliminary studies about effects of colostrum supplementation show its potential for increasing human exercise performance; however, more evidence across the lifespan is required to confirm effects and to understand mechanisms of action. The objectives are to determine the effect of 8 weeks of bovine colostrum supplementation, compared to whey protein supplementation on the following dependent variables in men and women 50 years and older while participating in a resistance-training program:

* muscle mass
* strength
* blood levels of growth factors and markers of inflammation
* urine levels of muscle and bone catabolic markers
* tests of cognitive ability It is hypothesized that bovine colostrum supplementation will result in greater increases in muscle mass, strength, blood IGF-1 levels (an anabolic hormone), and cognitive ability, and greater reductions in inflammation, and markers of muscle and bone catabolism, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 50 y or older

Exclusion Criteria:

* Milk allergies
* Contraindications to exercise as indicated by the Physical Activity Readiness Questionnaire

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
change from baseline in lean tissue mass at 8 weeks | baseline and 8 weeks
  Lean tissue mass assessed by dual energy x-ray absorptiometry
Change from baseline in Upper body strength at 8 weeks | baseline and 8 weeks
  Bench Press Strength
Change from baseline in Lower body strength at 8 weeks | baseline and 8 weeks
  Leg press strength

SECONDARY OUTCOMES:
Change from baseline in Insulin like growth factor-1 at 8 weeks | baseline and 8 weeks
  IGF-1 from serum
Change from baseline in upper body muscle thickness at 8 weeks | baseline and 8 weeks
  Muscle thickness of the elbow flexors assessed by ultrasound
Change from baseline in lower body muscle thickness at 8 weeks | baseline and 8 weeks
  Knee extensors muscle thickness assessed by ultrasound
Change from baseline in muscle catabolism at 8 weeks | baseline and 8 weeks
  Urinary 3-methylhistidine levels
Change from baseline in bone catabolism at 8 weeks | Baseline and 8 weeks
  Urinary cross-linked N-telopeptides of type I collagen
Number of Participants with Adverse Events as a Measure of Safety and Number of Participants with Adverse Events as a Measure of Safety and Tolerability | continuously throughout 8 weeks
  Adverse events collected on adverse event forms
Change from baseline in inflammation at 8 weeks | baseline and 8 weeks
  Serum cytokine markers of inflammation (IL-6 and TNF-alpha)
Change from baseline in cognitive ability at 8 weeks | baseline and 8 weeks
  The Telephone Interview of Cognitive Status

CONTACTS AND LOCATIONS:
Overall Officials: Philip D Chilibeck, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Antonio J, Sanders MS, Van Gammeren D. The effects of bovine colostrum supplementation on body composition and exercise performance in active men and women. Nutrition. 2001 Mar;17(3):243-7. doi: 10.1016/s0899-9007(00)00552-9. PMID 11312068
- [Background] Kerksick CM, Rasmussen C, Lancaster S, Starks M, Smith P, Melton C, Greenwood M, Almada A, Kreider R. Impact of differing protein sources and a creatine containing nutritional formula after 12 weeks of resistance training. Nutrition. 2007 Sep;23(9):647-56. doi: 10.1016/j.nut.2007.06.015. PMID 17679046